CLINICAL TRIAL: NCT04029896
Title: Individual Patient Expanded Access IND of Autologous Adipose-derived Mesenchymal Stem Cells for the Treatment of Cerebral Palsy
Brief Title: Individual Patient Expanded Access IND of Hope Biosciences Autologous Adipose-derived Mesenchymal Stem Cells for the Treatment of Cerebral Palsy
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBCP01
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: CP; stem cells; MSCs; spastic; paralysis; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Paralysis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — intravenous infusion of Hope Biosciences autologous adipose-derived stem cells

SUMMARY:
This is an Individual Patient Expanded Access Protocol of Autologous HB-adMSCs for the Treatment of Cerebral Palsy (CP) with the primary goal of treating 1 individual with CP who has exhausted all treatment options, his condition has not improved, his quality of life is severely affected by the condition and he has previously banked his mesenchymal stem cells. There are no FDA approved, fully restorative treatments for CP. The subject will receive 8 autologous HB-adMSC infusions of 50 million (50 x 10^6 cells) total cells. A protocol amendment to administer additional HB-adMSC infusions may be submitted for IRB/FDA for approval depending on the patient's response, AE/SAEs, and cell expansion characteristics.

DETAILED DESCRIPTION:
Once the eligibility is confirmed, approximately 1-3 weeks after the screening/baseline visit, the subject will return for the first infusions. Subsequent treatments will occur every other week.

On each of these visits, the subject will receive one autologous HB-adMSC infusion of 50 million (50 x 10^6 cells) total cells. Every infusion visit will include the following procedures:

1. Interval H&P update,
2. Weight
3. Vital signs monitoring (Heart Rate, BP, Resp., Temp., SpO2),
4. A urine and blood sample for clinical labs (CBC with diff., CMP, and Coagulation Panel, Serum Leptin),
5. A verification of patient/LAR consent will be verbally performed,
6. The HB-adMSC infusion will be given via IV over a 1 hour period.
7. The subject will then be monitored for a minimum of 4hr.
8. 24-hour telephone assessment for adverse events
9. Video Documentation

Follow Up Visits Week 4, 8, 12 and 16 (Safety Assessments)

The patient will be assessed for adverse events 24 hours after each infusion with a follow up phone call. 4 weeks after the first infusion have occurred, the subject will return to the clinical site for an onsite safety assessment, which will be repeated at week 8, 12, and 16. Each one of these on-site safety assessments will include:

1. Review and update medical history,
2. Update concomitant medications list
3. Video documentation
4. Weight
5. Vital signs (Heart Rate, BP, Respirations, Temp., SpO2),
6. Physical exam,
7. A urine and blood sample for clinical labs (CBC with diff., CMP, and Coagulation Panel and serum leptin)
8. SARAH assessment on Weeks 4, 12 and 16.
9. Adverse event monitoring Follow Up Visit Week 26 (Safety Assessments)

1. Review and update medical history, 2. Update concomitant medications list 3. Weight 4. Vital signs (Heart Rate, BP, Respirations, Temp., SpO2), 5. Physical exam, 6. A urine and blood sample for clinical labs (CBC with diff., CMP, and Coagulation Panel and serum leptin), 7. Brain MRI 8. The SARAH (motor-functional evaluation scale for children and adolescents with cerebral palsy) 9. Adverse event monitoring 10. Video documentation

Follow Up Visit Week 52 (Safety Assessments-End of Study)

1. Review and update medical history,
2. Update concomitant medications list
3. Weight
4. Vital signs (Heart Rate, BP, Respirations, Temp., SpO2),
5. Physical exam,
6. A urine and blood sample for clinical labs (CBC with diff., CMP, and Coagulation Panel and serum leptin),
7. Chest X ray (PA Single view)
8. The SARAH (motor-functional evaluation scale for children and adolescents with cerebral palsy)
9. Adverse event monitoring
10. Video documentation

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Cerebral Palsy
2. 3 years and older.

Exclusion Criteria:

1. Recent or ongoing infection
2. Clinically significant cardiovascular, lung, renal, hepatic, or endocrine disease.
3. Immunosuppression as defined by WBC < 3, 000 cells/ml at baseline screening.
4. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSC administration.
5. Participation in other interventional research studies.
6. Unwillingness to return for follow-up visits.

Min Age: 3 Years | Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

REFERENCES:
- See also: Hope Biosciences — http://www.hope.bio